CLINICAL TRIAL: NCT03551223
Title: Neural Damage and Anesthetic Treatment in the Preeclamptic Parturient; a Prospective Observational Cohort Study.
Brief Title: Neural Damage and Anesthetic Treatment in the Preeclamptic Parturient; a Prospective Observational Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0504-17
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-06

CONDITIONS: Phosphopyruvate Hydratase
MeSH Terms: interventions — Phosphopyruvate Hydratase; S100 Calcium Binding Protein beta Subunit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5 cc of venous blood will be drawn from each of the participants and will be assed for NSE and S100B serum levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women undergoing cesarean delivery with general anesthesia: Preeclamptic parturients undergoing cesarean delivery under general anesthesia
  Interventions: Biological: Neuron specific enolase (NSE)
- Women undergoing cesarean delivery with spinal anesth: Preeclamptic parturients undergoing cesarean delivery under regional-spinal anesthesia
  Interventions: Biological: Neuron specific enolase (NSE)

INTERVENTIONS:
Biological: Neuron specific enolase (NSE) — 5 cc of venous blood will be drawn from all of the participants and be examined for NSE and S100 B serum levels in order to evaluate evaluate which anesthetic method (general anesthesia versus spinal anesthesia) is associated with reduced neuronal injury in a preeclamptic parturients undergoing a cesarean section.
  Other Names: S100B Protein

SUMMARY:
Objectives: Our primary objective is to evaluate the effect of anesthetic method (general versus regional anesthesia) on neural outcomes in the preeclamptic population undergoing cesarean delivery. Secondary outcome is to examine the fetal cerebral outcomes associated with the anesthetic method.

Methodology: This prospective, observational study, will include 50 preeclamptic parturients undergoing cesarean section under general and regional anesthesia.

Neuron specific enolase and S100B Protein are neuronal injury biomarkers. Increased levels of these biomarkers in serum indicate neuron damage. Following enrollment venous blood will be drawn from the participants and assessed for NSE and S100B serum levels at the following points; Upon hospital admission and one day postpartum. Furthermore in order to evaluate fetal outcomes upon fetal delivery, umbilical cord blood will be examined for NSE and S100B.

Study significance: While spinal anesthesia is the preferred anesthetic method for the preeclamptic parturient undergoing cesarean delivery, it remains uncertain which anesthetic method is neuroprotective.

This study will be the first study, to our knowledge, to examine the effect of anesthetic method on neuronal outcomes for a parturient with preeclampsia undergoing cesarean delivery, by the use of noninvasive cerebral biomarkers.

DETAILED DESCRIPTION:
Scientific background:

Preeclampsia is an idiopathic maternal, multi organ, specific pregnancy disorder, associated with significant maternal and perinatal morbidity and mortality. Preeclampsia complicates approximately 2-8% of all pregnancies. The disorder is characterized by new-onset of hypertension and proteinuria developing after gestational week 20. While the pathogenesis of the disease remains not completely understood, a possible explanation is endothelial cell dysfunction in which placenta-derived mediators causes multisystem organ dysfunction .

Preeclampsia increases the risk for acute cerebrovascular complications such as intracerebral hemorrhage, cerebral edema and eclampsia. Treatment with magnesium sulfate reduces the risk for seizures and treatment with antihypertensive therapy reduces the risk for a stroke , however the only effective treatment for the syndrome is prompt delivery of the fetus .

When considering the optimal anesthetic method for a preeclamptic parturient undergoing cesarean delivery, neuraxial anesthetic techniques, when feasible, are strongly preferred to general anesthesia (GA) . Spinal anesthesia (SA) is favored over general anesthesia since it is associated with increased benefits and reduced risks compared with general anesthesia. Increased benefits of SA include higher patient satisfaction, decreased pain and favorable neonatal outcomes. GA has been associated with increased risk for aspiration, unstable hemodynamics and difficult airway management . In addition GA has been shown to increase the risk for a stroke in women with preeclampsia . Nevertheless GA is sometime used in the preeclamptic parturient due to maternal or fetal indications with an incidence as high as 44% in some European countries .

Accumulative evidence from animal studies indicate that general anesthetic agents are neurotoxic and can induce subsequent behavioral abnormalities in the developmental mind . However the fetal and pediatric implications remain inconclusive. In a population-based birth cohort study fetal exposure to general anesthesia during cesarean delivery was not associated with increased risk for learning disabilities compared to delivering vaginally . In contrast in a population-based birth cohort study conducted in Taiwan the incidence of autism was increased in neonates who were delivered by cesarean delivery under general anesthesia compared with regional anesthesia .

Despite experts favoring neuraxial anesthesia for the preeclamptic population, to date research remains inconclusive regarding which anesthetic method is neuroprotective.

In recent years numerous biochemical tests have become usual clinical cerebral damage biomarkers, amongst them is the Neuron specific enolase (NSE). The NSE is an intracytoplasmic glycolytic enzyme enolase . The enzyme is expressed in neurons and neuroendocrine tissue . Increased levels of NSE are released into the blood circulation according to the death rate of those cells . Elevated levels of NSE have been observed after severe head trauma and in association to postoperative cognitive dysfunction .

S100B Protein, an additional neuronal injury biomarker, is an acidic calcium-binding protein, and physiological serum levels of S100B protein are low . The protein is found primarily in astrocytes and Schwann cells and has both intracellular and extracellular targets.

Elevated serum and CSF levels of S100B indicate neural damage . Research evaluating cerebral damage biomarkers in parturients with preeclampsia has found increased levels of neuronal injury biomarkers compared with healthy parturients . Furthermore increased plasma levels of S100B have been correlated with neurological symptoms in the form of visual disturbances . Lisa et al demonstrated persistent increased levels of NSE up to one year postpartum .

Additionally, various studies have examined the correlation between cerebral biomarkers levels in umbilical cord blood, amniotic fluid and fetal pathological conditions: intra uterine fetal death, preterm delivery, cerebral palsy and preeclampsia . Tskitishvili, et al showed increased levels of cerebral injury damage in amniotic fluid of parturients with preeclampsia .

In this study we aim to evaluate the effect of anesthetic method on neural outcomes in the preeclamptic population undergoing cesarean delivery.

Specific Aims:

Our primary objective is to examine which anesthetic method (GA versus RA) is associated with reduced neural damage as measured by NSE and S100B serum levels in preeclamptic parturients undergoing cesarean delivery.

Our secondary objective is to examine the effect of anesthetic method on fetal cerebral outcomes as measured by NSE and S100B umbilical cord blood levels in parturients with preeclampsia.

Study Design:

This is a prospective, single center, observational trial to assess the effect of anesthetic method on cerebral outcomes. The study will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital.

Fifty preeclamptic parturients aged 18 and above, undergoing cesarean delivery under SA or GA, will be included in the study.

This study is a purely observational study, it will not have any clinical intervention nor will it interfere with standard cesarean delivery protocols in any way. Inclusion criteria Fifty preeclamptic parturients age 18 and above presenting for cesarean delivery under SA or GA, with ability to comply with study requirements will be enrolled in the study.

Exclusion criteria

The following parturients will be excluded:

1. Parturients under age 18
2. Parturients undergoing a vaginal delivery.
3. Parturients unable to sign an informed consent forum.

Study enrollment:

All preeclamptic parturients will be recruited upon admission to the women's emergency room. All participating patients will undergo an informed consent process, which will include a through explanation of the study design and patient requirements, by the study investigator. Following which patients will be requested to sign the informed consent document.

Index procedure:

Following obtaining approval from parturients 5 cc of venous blood will be drawn from each of the participants and will be examined for NSE and S100B serum levels at the following time points:

1. Upon hospital admission following obtaining informed consent approval.
2. Upon fetal delivery, umbilical cord blood will be examined for NSE and S100B.
3. 1 day postpartum. The blood samples will be collected in heparin containing tubes, the samples will be kept in room temperature for no longer than an hour before being sent to the laboratory for centrifugation. Following centrifugation the samples will be frozen at -70 °C until levels of NSE and S100B can be analyzed. Plasma levels will be tested to detect NSE and S100B levels using commercially available kits (Liasion Sangtec 100) according to the manufacturer's recommendations.

Intraoperative anesthetic technique will be administered at anesthesiologists' discretion. The study cohort will be divided into two groups: women undergoing cesarean delivery under general anesthesia, and women undergoing cesarean delivery under regional-spinal anesthesia.

NSE and S100B levels will be compared for both groups in order to evaluate which anesthetic method is associated with reduced neuronal injury Additionally, umbilical cord blood NSE and S100B levels will be compared for both groups, in order to assess the fetal outcomes of each anesthetic method.

Data collection:

For each participant the following additional data will be collected and documented:

1. Demographic data obstetric age, weight, height,
2. Obstetric data; gravidity and parity, obstetric history comorbidities, regular medication and preeclampsia management protocols and more.
3. Anesthetic and analgesic data: type of anesthesia / analgesia, anesthetic drug solution, anesthetic drug doses, vasopressor treatment, hemodynamic data, and other anesthetic data.

ELIGIBILITY:
Inclusion Criteria:

Fifty preeclamptic parturients age 18 and above presenting for cesarean delivery under SA or GA, with ability to comply with study requirements will be enrolled in the study.

Exclusion Criteria:

The following parturients will be excluded:

1. Parturients under age 18
2. Parturients undergoing a vaginal delivery.
3. Parturients unable to sign an informed consent forum.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Fifty preeclamptic parturients aged 18 and above, undergoing cesarean delivery under SA or GA, will be included in the study.
  This study is a purely observational study, it will not have any clinical intervention nor will it interfere with standard cesarean delivery protocols in any way.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
NSE serum levels | 1 Day postpartum
  Maternal serum NSE levels after delivery in both study groups
S100 B protein | 1 Day postpartum
  Maternal serum S100B levels after delivery in both study groups. Maternal serum NSE levels after delivery in both study groups

SECONDARY OUTCOMES:
Fetal serum NSE levels | At delivery
  Umbilical cord serum NSE levels
Fetal serum S100b levels | At delivery
  Umbilical cord serum S100b levels

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bergman L, Akerud H. Plasma Levels of the Cerebral Biomarker, Neuron-Specific Enolase, are Elevated During Pregnancy in Women Developing Preeclampsia. Reprod Sci. 2016 Mar;23(3):395-400. doi: 10.1177/1933719115604732. Epub 2015 Sep 8. PMID 26355117
- [Background] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Barry MJ, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Phillips WR, Phipps MG, Silverstein M, Simon MA, Tseng CW. Screening for Preeclampsia: US Preventive Services Task Force Recommendation Statement. JAMA. 2017 Apr 25;317(16):1661-1667. doi: 10.1001/jama.2017.3439. PMID 28444286
- [Background] Clark VA, Sharwood-Smith GH, Stewart AV. Ephedrine requirements are reduced during spinal anaesthesia for caesarean section in preeclampsia. Int J Obstet Anesth. 2005 Jan;14(1):9-13. doi: 10.1016/j.ijoa.2004.08.002. PMID 15627532
- [Background] Henke VG, Bateman BT, Leffert LR. Focused review: spinal anesthesia in severe preeclampsia. Anesth Analg. 2013 Sep;117(3):686-693. doi: 10.1213/ANE.0b013e31829eeef5. Epub 2013 Jul 18. PMID 23868886
- [Background] Tskitishvili E, Komoto Y, Temma-Asano K, Hayashi S, Kinugasa Y, Tsubouchi H, Song M, Kanagawa T, Shimoya K, Murata Y. S100B protein expression in the amnion and amniotic fluid in pregnancies complicated by pre-eclampsia. Mol Hum Reprod. 2006 Dec;12(12):755-61. doi: 10.1093/molehr/gal083. Epub 2006 Oct 5. PMID 17023485
- [Background] Huang CJ, Fan YC, Tsai PS. Differential impacts of modes of anaesthesia on the risk of stroke among preeclamptic women who undergo Caesarean delivery: a population-based study. Br J Anaesth. 2010 Dec;105(6):818-26. doi: 10.1093/bja/aeq266. Epub 2010 Oct 6. PMID 20926478
- [Background] Pant M, Fong R, Scavone B. Prevention of peri-induction hypertension in preeclamptic patients: a focused review. Anesth Analg. 2014 Dec;119(6):1350-6. doi: 10.1213/ANE.0000000000000424. PMID 25405694
- [Background] De Tina A, Palanisamy A. General Anesthesia During the Third Trimester: Any Link to Neurocognitive Outcomes? Anesthesiol Clin. 2017 Mar;35(1):69-80. doi: 10.1016/j.anclin.2016.09.007. Epub 2016 Dec 12. PMID 28131121
- [Background] Graham MR. Clinical update regarding general anesthesia-associated neurotoxicity in infants and children. Curr Opin Anaesthesiol. 2017 Dec;30(6):682-687. doi: 10.1097/ACO.0000000000000520. PMID 28915132
- [Background] Sprung J, Flick RP, Wilder RT, Katusic SK, Pike TL, Dingli M, Gleich SJ, Schroeder DR, Barbaresi WJ, Hanson AC, Warner DO. Anesthesia for cesarean delivery and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Aug;111(2):302-10. doi: 10.1097/ALN.0b013e3181adf481. PMID 19602960
- [Background] Chien LN, Lin HC, Shao YH, Chiou ST, Chiou HY. Risk of autism associated with general anesthesia during cesarean delivery: a population-based birth-cohort analysis. J Autism Dev Disord. 2015 Apr;45(4):932-42. doi: 10.1007/s10803-014-2247-y. PMID 25256350
- [Background] Lee A, Kim SH, Hong JY, Hwang JH. Effect of anesthetic methods on cerebral oxygen saturation in elderly surgical patients: prospective, randomized, observational study. World J Surg. 2012 Oct;36(10):2328-34. doi: 10.1007/s00268-012-1676-z. PMID 22736340
- [Background] Hoppenstein D, Zohar E, Ramaty E, Shabat S, Fredman B. The effects of general vs spinal anesthesia on frontal cerebral oxygen saturation in geriatric patients undergoing emergency surgical fixation of the neck of femur. J Clin Anesth. 2005 Sep;17(6):431-8. doi: 10.1016/j.jclinane.2004.09.013. PMID 16171663
- [Background] Hirose N, Kondo Y, Maeda T, Suzuki T, Yoshino A. Relationship between regional cerebral blood volume and oxygenation and blood pressure during spinal anesthesia in women undergoing cesarean section. J Anesth. 2016 Aug;30(4):603-9. doi: 10.1007/s00540-016-2165-6. Epub 2016 Mar 24. PMID 27011334
- [Background] Sun S, Liu NH, Huang SQ. Role of cerebral oxygenation for prediction of hypotension after spinal anesthesia for caesarean section. J Clin Monit Comput. 2016 Aug;30(4):417-21. doi: 10.1007/s10877-015-9733-4. Epub 2015 Jul 18. PMID 26186992
- [Background] Trakas E, Domnina Y, Panigrahy A, Baust T, Callahan PM, Morell VO, Munoz R, Bell MJ, Sanchez-de-Toledo J. Serum Neuronal Biomarkers in Neonates With Congenital Heart Disease Undergoing Cardiac Surgery. Pediatr Neurol. 2017 Jul;72:56-61. doi: 10.1016/j.pediatrneurol.2017.04.011. Epub 2017 Apr 21. PMID 28571730
- [Background] van Munster BC, Korse CM, de Rooij SE, Bonfrer JM, Zwinderman AH, Korevaar JC. Markers of cerebral damage during delirium in elderly patients with hip fracture. BMC Neurol. 2009 May 27;9:21. doi: 10.1186/1471-2377-9-21. PMID 19473521
- [Background] Tomaszewski D. Biomarkers of Brain Damage and Postoperative Cognitive Disorders in Orthopedic Patients: An Update. Biomed Res Int. 2015;2015:402959. doi: 10.1155/2015/402959. Epub 2015 Aug 31. PMID 26417595
- [Background] Georgiadis D, Berger A, Kowatschev E, Lautenschlager C, Borner A, Lindner A, Schulte-Mattler W, Zerkowski HR, Zierz S, Deufel T. Predictive value of S-100beta and neuron-specific enolase serum levels for adverse neurologic outcome after cardiac surgery. J Thorac Cardiovasc Surg. 2000 Jan;119(1):138-47. doi: 10.1016/s0022-5223(00)70229-7. PMID 10612773
- [Background] Wikstrom AK, Ekegren L, Karlsson M, Wikstrom J, Bergenheim M, Akerud H. Plasma levels of S100B during pregnancy in women developing pre-eclampsia. Pregnancy Hypertens. 2012 Oct;2(4):398-402. doi: 10.1016/j.preghy.2012.03.001. Epub 2012 Mar 16. PMID 26105610
- [Background] Vettorazzi J, Torres FV, de Avila TT, Martins-Costa SH, Souza DO, Portela LV, Ramos JG. Serum S100B in pregnancy complicated by preeclampsia: A case-control study. Pregnancy Hypertens. 2012 Apr;2(2):101-5. doi: 10.1016/j.preghy.2011.11.004. Epub 2011 Dec 13. PMID 26105095
- [Background] Bergman L, Akerud H, Wikstrom AK, Larsson M, Naessen T, Akhter T. Cerebral Biomarkers in Women With Preeclampsia Are Still Elevated 1 Year Postpartum. Am J Hypertens. 2016 Dec 1;29(12):1374-1379. doi: 10.1093/ajh/hpw097. PMID 27653032
- [Background] Gazzolo D, Vinesi P, Marinoni E, Di Iorio R, Marras M, Lituania M, Bruschettini P, Michetti F. S100B protein concentrations in cord blood: correlations with gestational age in term and preterm deliveries. Clin Chem. 2000 Jul;46(7):998-1000. No abstract available. PMID 10894846
- [Background] Lu H, Huang W, Chen X, Wang Q, Zhang Q, Chang M. Relationship between premature brain injury and multiple biomarkers in cord blood and amniotic fluid. J Matern Fetal Neonatal Med. 2018 Nov;31(21):2898-2904. doi: 10.1080/14767058.2017.1359532. Epub 2017 Aug 3. PMID 28738706